CLINICAL TRIAL: NCT05700786
Title: Mindful Compassion for Perfectionism: A Waiting-list Randomized Controlled Trial
Brief Title: Mindful Compassion for Perfectionism
Acronym: MCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tages Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCP-2022
Record Dates: First submitted 2022-03-11; First posted 2023-01-26 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Perfectionism
Keywords: perfectionism; mindfulness; self-criticism; group psychotherapy

STUDY DESIGN:
Intervention Model Description: Pragmatic waiting-list randomized controlled trial with blinded outcome assessment
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study design reflects an external, third-party evaluation. The evaluation team (i.e. the researcers conducting the analysis) will be independent from both the application vendor (i.e. the therapists conducting the intervention) and the recruitment team (i.e. the researchers recruiting and randomly allocating the participants).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The control group is made up of participants who are eligible but not assigned to the treatment. For ethical reasons they will be able to access the intervention once the experimental group has concluded the study. During the waiting-list phase, participants can access a mental health intervention, but in this case they are excluded from the study. Participants are told that there is only one possible active group and therefore a waiting-list is created. This explanation is given to reduce a worsening symptom bias for feeling "excluded" from treatment.
- Experimental Group 1 - Online Format (Active Comparator): The experimental intervention is an integrative mindful compassion group therapy as manualized by Cheli, Cavalletti, Flett & Hewitt (2020). The structure was outlined on the base of standard mindfulness-based interventions, comprising eight 2-hour online group sessions and one day of silence lasting 4 hours. The contents and the phases of the intervention were rooted in two different frameworks. On the one hand, the sequence of and the types of practices were defined in accordance with the mindful compassion protocol (Gilbert & Choden, 2014). On the other hand, the shared conceptualization of perfectionism and its role in triggering, maintaining, and inducing relapses in personality disoders was proposed through the relational model by Hewitt and colleagues (2017). The hybrid format (online weekly sessions plus an in presence half-day of silence) has been developed in accordance with existing COViD-19 emergency and rules.
  Interventions: Behavioral: Mindful compassion for perfectionism
- Experimental Group 2 - Online Format (Active Comparator): The experimental intervention is an integrative mindful compassion group therapy as manualized by Cheli, Cavalletti, Flett & Hewitt (2020). The structure was outlined on the base of standard mindfulness-based interventions, comprising eight 2-hour in presence group sessions and one day of silence lasting 4 hours in presence. The contents and the phases of the intervention were rooted in two different frameworks. On the one hand, the sequence of and the types of practices were defined in accordance with the mindful compassion protocol (Gilbert & Choden, 2014). On the other hand, the shared conceptualization of perfectionism and its role in triggering, maintaining, and inducing relapses in personality disoders was proposed through the relational model by Hewitt and colleagues (2017).
  Interventions: Behavioral: Mindful compassion for perfectionism

INTERVENTIONS:
Behavioral: Mindful compassion for perfectionism — The intervention is a 8-week group psychotherapy in a hybrid format: 8 weekly online sessions lasting 2 hours plus an in presence half-day of silence lasting 4 hours.
  Arms: Experimental Group 1 - Online Format; Experimental Group 2 - Online Format

SUMMARY:
The aim of this study is to confirm the feasibility of an integrative form of group psychotherapy in treating perfectionism. In a previous pilot study we suggested that this new treatment is safe and feasible, also reporting a significant reduction of perfectionism at final assessment. The intervention integrates the Paul Hewitt relational model of perfectionism and the Paul Gilbert Compassion Focused Therapy. We will explore the feasibility of the proposed group therapy through a three-arm waiting-list randomized controlled trial. Our hypothesis is that those in the treatment groups (either online or in presence format) will show at the end of the intervention a lower level of perfectionsm than those in the control group.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all partecipants giving written informed consent will undergo a psychological assessment so as to determine eligibility for study entry. Patients who meet the eligibility requirements will be randomized in a double-blind manner in a 1:1 ratio to (i) new integrative group psychotherapy through an in presence format, (ii) the same integrative group psychotherapy through an online format, (iii) a waiting-list control group. At the end of active experimental groups treatment (2 months), all the partecipants will have access to the final follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 18 and 30
* Reporting at least a clinically significant value at Multidimensional Perfectionsm Scale (at least one of the dimensions must have scores equal to or greater than the clinical population mean of the questionnaire manual)

Exclusion Criteria:

* Being diagnosed with neurodevelopmental or schizophrenia/psychosis spetrum disoders;
* Being under either psychiatric or psychological treatment

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Feasibility (adverse events; adherence) | 2 measurements: one at baseline assessment; one at final assessment. Initial assessment will be 1 month priori the intervention, the final assessment at the end of the intervention (2 months after the beginning of the intervention).
  Feasibility is defined on the basis of two criteria: absence of adverse events (i.e. dropouts; hospitalization; etc.) and adequate adherence (i.e. maximum 1 skipped session per participant)
Betwen-groups effectiveness (perfectionism) | 2 measurements: one at baseline assessment; one at final assessment. Initial assessment will be 1 month priori the intervention, the final assessment at the end of the intervention (2 months after the beginning of the intervention).
  At the final assessment, the experimental group's Perfectionistic Cognitions Inventory (PCI) scores are significantly lower than those of the control group (the differences in the initial assessment must be insignificant). Higher scores of PCI (ranging between 0 to 100) are indicative of higher perfectionistic worry

SECONDARY OUTCOMES:
Withing-group effectiveness (perfectionism) | 2 measurements: one at baseline assessment; one at final assessment. Initial assessment will be 1 month priori the intervention, the final assessment at the end of the intervention (2 months after the beginning of the intervention).
  In the experimental group the scores on the Perfectionistic Cognitions Inventory (PCI) must show a significant difference between initial and final assessment. Higher scores of PCI (ranging between 0 to 100) are indicative of higher perfectionistic worry

CONTACTS AND LOCATIONS:
Overall Officials: Simone Cheli, PhD, Principal Investigator — Tages Onlus; Paul L Hewitt, PhD, Study Chair — British Columbia University; Gil Goldzweig, PhD, Study Chair — The Academic College of Tel-Aviv Yaffo
Locations (1):
- Centro di Psicologia e Psicoterapia Tages Onlus - Firenze, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be made available at the beginning of the active treatment phase and the raw data at the end of the study. All information will be uploaded to the Open Science Foundation.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol, SAP, ICF and CSR will be available before the end of February 2023
Access Criteria: All material will be freely accessible to anyone on the Open Science Foundation (see link below).
URL: https://osf.io/46p3s/?view_only=4f7ec72f10714959af0936457ac80e85

REFERENCES:
- [Background] Cheli S, Cavalletti V, Flett GL, Hewitt PL. Mindful compassion for perfectionism in personality disorders: A pilot acceptability and feasibility study. BPA - Applied Psychology Bulletin (Bollettino di Psicologia Applicata). 2020; 68(287): 55-65. https://doi.org/10.26387/bpa.287.5
- [Background] Hewitt PL, Mikail SF, Dang SS, Kealy D, Flett GL. Dynamic-relational treatment of perfectionism: An illustrative case study. J Clin Psychol. 2020 Nov;76(11):2028-2040. doi: 10.1002/jclp.23040. Epub 2020 Aug 15. PMID 33245562
- [Background] Hewitt PL, Qiu T, Flynn CA, Flett GL, Wiebe SA, Tasca GA, Mikail SF. Dynamic-relational group treatment for perfectionism: Informant ratings of patient change. Psychotherapy (Chic). 2020 Jun;57(2):197-205. doi: 10.1037/pst0000229. Epub 2019 May 20. PMID 31107049
- [Background] Hewitt PL, Smith MM, Deng X, Chen C, Ko A, Flett GL, Paterson RJ. The perniciousness of perfectionism in group therapy for depression: A test of the perfectionism social disconnection model. Psychotherapy (Chic). 2020 Jun;57(2):206-218. doi: 10.1037/pst0000281. Epub 2020 Jan 30. PMID 31999191
- [Background] Smith MM, Sherry SB, Ray C, Hewitt PL, Flett GL. Is perfectionism a vulnerability factor for depressive symptoms, a complication of depressive symptoms, or both? A meta-analytic test of 67 longitudinal studies. Clin Psychol Rev. 2021 Mar;84:101982. doi: 10.1016/j.cpr.2021.101982. Epub 2021 Jan 26. PMID 33556805
- [Background] Gilbert P. Compassion: From Its Evolution to a Psychotherapy. Front Psychol. 2020 Dec 9;11:586161. doi: 10.3389/fpsyg.2020.586161. eCollection 2020. PMID 33362650
- [Background] Gilbert P. Evolution and depression: issues and implications. Psychol Med. 2006 Mar;36(3):287-97. doi: 10.1017/S0033291705006112. Epub 2005 Oct 20. PMID 16236231
- [Background] Petrocchi N, Dentale F, Gilbert P. Self-reassurance, not self-esteem, serves as a buffer between self-criticism and depressive symptoms. Psychol Psychother. 2019 Sep;92(3):394-406. doi: 10.1111/papt.12186. Epub 2018 Jun 15. PMID 29907988
- [Background] McEwan K, Gilbert P. A pilot feasibility study exploring the practising of compassionate imagery exercises in a nonclinical population. Psychol Psychother. 2016 Jun;89(2):239-43. doi: 10.1111/papt.12078. Epub 2015 Oct 10. PMID 26454144
- [Background] GILBERT, P. & CHODEN, K. (2014). Mindful compassion: How the science of compassion can help you understand your emotions, live in the present, and connect deeply with others. New Harbinger Publications.
- [Background] HEWITT, P.L., FLETT, G.L. & MIKAIL, S.F. (2017). Perfectionism: A relational approach to conceptualization, assessment, and treatment. New York:The Guilford Press.